CLINICAL TRIAL: NCT02939924
Title: Prospective, Multi-Center, Open, Single Arm Study for the Treatment of Patients Presenting De Novo Lesions in the Superficial Femoral and/or Popliteal Arteries Using a Kanshas Drug Coated Balloon Catheter.
Brief Title: Treatment of Patients With Lesions in the Superficial Femoral and/ or Popliteal Arteries Using Kanshas Paclitaxel-coated Balloon Catheter.
Acronym: KANSHAS-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T129E4
Record Dates: First submitted 2016-10-17; First posted 2016-10-20 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2023-09

CONDITIONS: Femoropopliteal Occlusive Disease; Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DCB treatment (Experimental): Patient treated with Kanshas DCB
  Interventions: Device: Kanshas DCB

INTERVENTIONS:
Device: Kanshas DCB — The appropriate Kanshas DCB size is selected after review of the patient's baseline angiogram and determination of the reference vessel diameter and lesion length. The balloons is sized to ensure the full length of the lesion is treated. The initial inflation of the study device should be approximately 1 minute for optimal drug release. In order to optimize lesion dilatation, longer inflation times are possible at the discretion of the operator.

SUMMARY:
Assessing the safety and effectiveness of the Kanshas Paclitaxel-coated Balloon Catheter in the treatment of de novo lesions in the superficial femoral (SFA) and/or popliteal arteries.

DETAILED DESCRIPTION:
The KANSHAS 1 (K-1) trial investigates the inhibition of restenosis using the Kanshas Paclitaxel-coated Balloon Catheter in the treatment of de novo lesions in the superficial femoral and/or popliteal arteries.

This clinical study is a prospective, multi-center, open, single-arm study. Up to 50 patients will be enrolled at 2 sites in Belgium and 4 sites in Germany. Follow-ups are scheduled before discharge, at 1 month (Clinic Visit or Phone FU), 6 months, 1-year, 2-years (Clinic Visits), 3-, 4- and 5- years (Clinic Visits or Phone FU).

Primary outcome measure:

* freedom from device-and procedure-related death through 30 days.
* freedom from target limb amputations and clinically driven target lesion revascularization through 6 months.

ELIGIBILITY:
Inclusion Criteria:

General:

1. Clinically significant symptomatic leg ischemia, requiring treatment of the SFA and/or popliteal artery;
2. Able and willing to provide informed consent prior to study procedures;
3. Able and willing to comply with follow-up requirements;
4. Rutherford Clinical Category of 2-4;
5. Resting ABI of <0.9 or abnormal exercise ABI;
6. ≥18 years old;
7. Life expectancy is >2 year;

   Angiographic Criteria:
8. Cumulative lesion length ≥4 and ≤15 cm within the target vessel; Cumulative lesion consists of either a single de novo lesion or multiple lesions within the 4-15 cm segment; multiple lesions require to meet all the following;

   * Separated by a gap of ≤ 3 cm;
   * Able to be treated as a single lesion;
   * Total combined lesion length including 3cm gap meets requirements;
9. Lesion location starts ≥2 cm distal to the common femoral bifurcation and terminates at ≥2 cm proximal to the origin of the tibio-peroneal trunk;
10. Clinically and hemodynamically significant de novo stenosis (>70% stenosis by visual estimate) or occlusion;
11. Target vessel diameter between ≥4 and ≤6 mm and able to be treated with available device size matrix;
12. Successful, uncomplicated (without use of a crossing device) antegrade wire crossing of lesion;
13. A patent inflow artery free from significant lesion (≥50% stenosis) as confirmed by angiography (treatment of target lesion acceptable after successful treatment of ipsilateral iliac lesions); NOTE: Successful ipsilateral iliac artery treatment is defined as attainment of residual diameter stenosis ≤30% without death or major vascular complication.
14. At least one patent native outflow artery to the ankle, free from significant (≥50%) stenosis as confirmed by angiography that has not previously been revascularized;

Exclusion Criteria:

1. Pregnant or lactating females;
2. Co-existing clinically significant aneurismal disease of the abdominal aorta, iliac or popliteal arteries;
3. Significant gastrointestinal bleeding or any coagulopathy that would contraindicate the use of anti-platelet therapy;
4. Known intolerance to study medications, paclitaxel or contrast agents;
5. Patient participating in another investigational device or drug study that has not reached the primary endpoint;
6. History of hemorrhagic stroke within 2 months;
7. Previous or planned surgical or interventional procedure within 30 days of the study procedure;
8. Diagnosed liver failure, renal failure, chronic kidney disease, unstable angina pectoris, or myocardial infarction within 30 days of the procedure;
9. Presence of significant stenosis or occlusion of the inflow tract that cannot be successfully treated prior to study consideration. Successful is defined as <30% residual stenosis of ipsilateral iliac artery with no major complications;
10. Acute thrombus in target vessel;
11. At site of target lesion, use of adjunctive therapies (i.e. laser, atherectomy, cryoplasty, scoring/cutting balloon, brachytherapy);
12. Outflow arteries (distal popliteal, anterior or posterior tibial or peroneal arteries) with significant lesions (≥50% stenosis) may not be treated during the same procedure;
13. Has in-stent restenosis in the target lesion;
14. Previous treatment with a drug coated PTA balloon catheter or drug eluting stent in the target vessel within 12 months of the index procedure;
15. Previous peripheral bypass affecting the target limb;
16. Has injuries in the target vessel, such as major flow-limiting dissection ( > NHLBI Grade C) and perforation, requiring stenting prior to enrollment;
17. Obvious subintimal recanalization or intentional subintimal recanalization in the occlusive lesions;
18. Presence of severe calcification in the target lesions that precludes endovascular treatment. Severe calcification is defined as circumferential calcification involving ≥ 50% of vessel diameter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of the study is a composite of freedom from device and procedure related deaths through 30 days, freedom from target limb amputation, and clinically driven target lesion revascularization (TLR) through 6 months. | 6 months
  Clinically-driven target lesion revascularization is defined as a restenosis of 50% or more in the target lesion with worsening symptoms, OR more as 70% stenosis without symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lichtenberg, MD, Principal Investigator — Karolinen-Hospital Klinikum Arnsberg, Germany
Locations (6):
- Belgium (2):
  - AZ Imelda, Bonheiden
  - AZ Sint Blasius, Dendermonde
- Germany (4):
  - Klinikum Hochsauerland Gmbh, Arnsberg
  - Uni-Herzzentrum, Bad Krozingen
  - Ev Luth Diakonissenanstalt, Flensburg
  - RoMed Klinikum, Rosenheim

IPD SHARING:
Plan to Share IPD: No